CLINICAL TRIAL: NCT04007172
Title: Effectiveness of Neural Therapy in Patients With Fibromiyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Tuğba Atan, Assoc. Prof., Hitit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-114
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Fibromyalgia
Keywords: neural therapy; physical theraphy; lidocain injection
MeSH Terms: conditions — Fibromyalgia | interventions — Anesthesia, Local; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural Therapy & home exercise program (Experimental): Intracutaneous quaddle injections were performed using 1% lidocaine preparation as a local anesthetic for local application to painful points with palpation on the back and shoulders and for the segmental application, 2 cm lateral to the midline of the C1-T5 vertebrae and on spinous processes.
  Both the groups received education about fibromyalgia and home exercise program, which included stretching, strengthening, and aerobic exercises.
  Interventions: Procedure: neural therapy
- Physical Therapy & home exercise program (Experimental): Physical therapy program was consist of transcutaneous electrical nerve stimulation- TENS (30-40 Hz, 20 minutes), hotpack (20 minutes) and continuous ultrasound (1mHz, 1.5w / cm2, 10 minutes) on painful points with palpation on the back and shoulders.
  Both the groups received education about fibromyalgia and home exercise program, which included stretching, strengthening, and aerobic exercises.
  Interventions: Device: Physical Therapy

INTERVENTIONS:
Procedure: neural therapy — Intracutaneous quaddle injections were performed using 1% lidocaine preparation as a local anesthetic for local application to painful points with palpation on the back and shoulders and for the segmental application, 2 cm lateral to the midline of the C1-T5 vertebrae and on spinous processes.
  Arms: Neural Therapy & home exercise program
Device: Physical Therapy — Physical therapy program was consist of transcutaneous electrical nerve stimulation- TENS (30-40 Hz, 20 minutes), hotpack (20 minutes) and continuous ultrasound (1mHz, 1.5w / cm2, 10 minutes) on painful points with palpation on the back and shoulders.
  Arms: Physical Therapy & home exercise program

SUMMARY:
Neural therapy is a regulation therapy that tries to correct this underlying autonomic dysfunction. In neural therapy; local painful areas, trigger points and symptomatic segments are included in the injection using local anesthetics and the underlying disruptive areas are investigated and treated. The aim of this study was to investigate the efficacy of neural therapy in fibromyalgia syndrome which is thought to have a neuroendocrine dysregulation disorder.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic disease characterized by widespread body pain, fatigue, sleep disturbance, and tenderness on palpation at trigger points in the musculoskeletal system.

Fibromyalgia prevalence is reported between 3% and 9%, and is three times more common in women than men. Although pharmacological and non-pharmacological approaches play a role in the treatment of the disease, the interest in non-pharmacological therapies has recently increased. In several studies, it has been shown that almost every fibromyalgia patient has applied at least one alternative and complementary medicine method such as Qigong, Tai Chi, yoga, mind body interventions, acupuncture, hydrotherapy, balneotherapy or phytotherapy.

Neural therapy is a regulation therapy that tries to correct this underlying autonomic dysfunction. In neural therapy; local painful areas, trigger points and symptomatic segments are included in the injection using local anesthetics and the underlying disruptive areas are investigated and treated. The aim of this study was to investigate the efficacy of neural therapy in fibromyalgia syndrome which is thought to have a neuroendocrine dysregulation disorder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed according to the American College of Rheumatology 2016 diagnostic criteria for fibromyalgia.

Exclusion Criteria:

* History of comorbid inflammatory rheumatic/ connective tissue diseases
* History of cardiovascular or musculoskeletal problems that could prevent them to participate in an exercise program

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female sex
Enrollment: 60 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Visual analog scale for pain | 4 weeks
  Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity.

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire | 4 weeks
  The Fibromyalgia Impact Questionnaire was designed to measure the health status of patients with fibromyalgia that contains the dimensions physical functioning (11 items), well-being (1 item), work situation (2 items), pain (1 item), fatigue /sleep (2 items), stiffness (2 items) and psychological symptoms (2 items). Total score range from 0 to 100, with higher scores indicating higher levels of symptoms and severity.
Short- form health survey 36 scores | 4 weeks
  Short- form health survey 36 contains 36 items which are used to evaluate the quality of life of patients with chronic pain. It measures eight different domains that address physical functioning, physical role limitation, pain, general health, vitality, social functioning, emotional role limitation and mental health. The score of each domain ranges from 0 (worse quality of life) to 100 (best quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğba Atan, Çorum, Turkey (Türkiye)